CLINICAL TRIAL: NCT01459731
Title: Optical Coherence Tomography Data Collection Study
Brief Title: Optical Coherence Tomography (OCT) Data Collection Study
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: OCT 200-47091
Record Dates: First submitted 2011-10-23; First posted 2011-10-26 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: No Eye Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Age 18-29
- Age 30-39
- Age 40-49
- Age 50-59
- Age 60-69
- Age 70+

SUMMARY:
Collect OCT data to evaluate the range and age trend of eye measurements.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able and willing to provide consent
* Able and willing to complete the required examininations and visit
* Refractive error within 8 diopters sphere and within 2 diopters cylinder in each eye
* Best corrected visual acuity of 20/30 or better in each eye

Exclusion Criteria:

* History of leukemia, AIDS, dementia or multiple sclerosis
* Concomitant use of hydroxycloroquine or chloroquine
* Family history of glaucoma among first degree relatives
* Intraocular pressure of 22mm Hg or greater in either eye
* Unreliable or abnormal visual field
* Active ocular disease
* Previously diagnosed with glaucoma or glaucoma suspect
* Congenital ocular abnormalities
* Previous intra-ocular surgery or laser treatment (other than refractive surgery or uncomplicated cataract surgery greater than 6 months previously)
* Anatomic narrow angle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No eye disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
range of eye measurements | Day 1

SECONDARY OUTCOMES:
age trend of eye measurements | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: George Comer, OD, MBA, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University; Michael Chaglasian, OD, Principal Investigator — Illinois Eye Institute; Jorge Cuadros, OD, PhD, Principal Investigator — Buena Vista Eye Care; David Garway-Heath, MD, Principal Investigator — Institute of Ophthalmology, University College London; Pinakin G Davey, OD, PhD, Principal Investigator — Western University of Health Sciences
Locations (5):
- United States (4):
  - Southern California College of Optometry, Fullerton, California
  - College of Optometry, Western University of Health Sciences, Pomona, California
  - Buena Vista Eye Care, San Jose, California
  - Illinois Eye Institute, Chicago, Illinois
- Institute of Ophthalmology, University College London, London, England, United Kingdom